CLINICAL TRIAL: NCT06287710
Title: Fluid Responsiveness Evaluation by a Non-invasive Method in Children, Extended to PREterm Infants - FRENCH-PREMA
Acronym: FRENCH-PREMA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/32
Record Dates: First submitted 2024-01-18; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Premature Baby 26 to 32 Weeks; Premature Baby 33 to 36 Weeks
Keywords: Circulatory failure (shock); volume expansion; echocardiography; Shock; goal-directed fluid management; preterm infants
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study of diagnostic accuracy: Patients included in this study would have received fluid expansion in all cases, as the prescription of 10 to 20ml/kg fluid expansion by the physician in charge is the main inclusion criterion.
  Interventions: Procedure: Non interventional study (study of diagnostic accuracy with an extra echocardiographic assessment).

INTERVENTIONS:
Procedure: Non interventional study (study of diagnostic accuracy with an extra echocardiographic assessment). — Study of diagnostic accuracy (non-interventional, prospective, monocentric). Fluid expansion will be delayed for a few minutes while our index test is performed. After fluid expansion, patient will undergo an echocardiographic assessment of response to fluid expansion (gold-standard test). This will allow to test the diagnostic performance of the index test for the "prediction" of fluid responsiveness.
  The index test is the ΔSVi-AC: indexed percentage of stroke volume variation between baseline and during a standardized abdominal compression. Stroke volume will be assessed by transthoracic echocardiography.
  Patient will undergo 3 echocardiographic assessment: At baseline (stroke volume, cardiac output, left ventricular ejection fraction), During a standardized abdominal compression (stroke volume),After the 10 to 20ml/kg fluid expansion prescribed by the physician in charge (cardiac output).

SUMMARY:
In this study, the investigators aim to validate a non-invasive marker of fluid-responsiveness in preterm infants (term below 37 gestational week) with acute circulatory failure based on standardized abdominal compression. This would allow physicians to identify which patient could benefit from a fluid expansion, thus avoiding a potentially useless or even dangerous fluid expansion, leading to fluid overload. To this end, the investigators will evaluate the diagnostic accuracy (sensitivity and specificity) of stroke volume variation induced by standardized abdominal compression for the diagnosis of fluid responsiveness (based on the gold-standard test: significant increase in cardiac index after fluid expansion).

DETAILED DESCRIPTION:
Fluid expansion is the cornerstone of acute circulatory failure treatment in children and preterm infants with acute circulatory failure. Although this therapy drastically reduced mortality, several studies in recent years have highlighted the adverse effects of excessive fluid expansion especially for preterm infants such as PDA, chronic lung disease and mortality. Currently, the search for indicators to predict fluid responsiveness is a major issue in neonatal intensive care. These indicators are based on Franck-Starling's law: if small changes in preload lead to an increase in cardiac output, then fluid responsiveness can be expected. However, in children, the only validated indicator (respiratory variability of peak aortic velocity) can only be used in the absence of any spontaneous respiratory movement, a rare situation in practice. Recently, two pediatric studies investigated a simple clinical test: hepatic or abdominal compression. This clinical maneuver, by increasing venous return via mobilization of the hepato-splanchnic reserve, induces a transient and reversible preload increase. The evaluation of the hemodynamic effects of this "endogenous fluid expansion" allowed, according to the authors, to accurately predict fluid responsiveness. However, several factors reduce the applicability of these results: the small number of studies on this subject, the smaller volume of fluid used than in clinical practice, and the population studied, composed almost exclusively of children in postoperative of cardiac surgery.

Thus, there is a need of reliable preloads markers to guide intravenous volume rescusitation in neonates.

In this study, the investigators will evaluate the diagnostic accuracy of abdominal compression for the diagnosis of fluid responsiveness in preterm infants (<37WA) with acute circulatory failure, hospitalized in neonatal intensive care unit for a medical or a non-cardiac surgical condition, for whom a fluid expansion was prescribed by the physician in charge. The index test will be the stroke volume variation following a standardized abdominal compression (before fluid expansion). The gold standard test will be the variation of cardiac output between baseline and after fluid expansion, a variation > 15% defining fluid responsiveness.

In this non interventional study of diagnostic accuracy, patients will undergo an extra echocardiographic assessment, but no supplemental blood test or invasive parameters will be collected. Simple clinical parameters will be collected within 4 hours after the fluid expansion.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn under 37 weeks of amenorrhea hospitalized in neonatal intensive care
* Prescription of a 10 to 20ml/kg fluid expansion (crystalloid, blood products or albumin) by the physician in charge, whose goal would be to increase cardiac output (based on clinical, biological and/or echographic criteria).

Exclusion Criteria:

* Acute cardiogenic pulmonary edema
* Hemodynamic instability making the delay necessary for abdominal compression and ultrasonography dangerous for the patient
* Non corrected congenital cardiopathy, or inferior to 15 days postoperative. Intra-abdominal hypertension or painful abdominal palpation
* Abdominal surgery in the last 15 days
* Supine position contraindicated or deleterious
* No investigator available to assess ultrasonographic measures
* Impairment of echocardiographic acoustic window or restless patient making ultrasonography impossible

Ages: 1 Minute to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: As this is a pilot study in a population of premature infants (term bellow 37 weeks of amenorrhea), the projected number of patients included will be 20, based on the department's active patient file, in order to have a minimum of 40 fluid expansion required for the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-11-17 (Estimated); Study Completion 2025-04-17 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy (sensitivity, specificity, positive predictive value, negative predictive value) of the index test (ΔSVi-AC) for the diagnosis of fluid responsiveness, | after abdominal compression, 30 minutes to 4 hours after baseline
  Diagnostic accuracy (sensitivity, specificity, positive predictive value, negative predictive value) of the index test (ΔSVi-AC) for the diagnosis of fluid responsiveness, defined by an increase of cardiac output > 15% after fluid expansion (ΔCO-FE > 15%, gold-standard test) Index test (ΔSVi-AC) will be calculated as the difference between SV after abdominal compression and SV at baseline, divided by SV at baseline (%). SV will be measured by echocardiographic assessment.
  Gold-standard test (ΔCO-FE) will be calculated as the difference between CO after fluid expansion and CO at baseline, divided by CO at baseline (%). CO will be measured by echocardiographic assessment.
  value) of the index test (ΔSVi-AC) for the diagnosis of fluid responsiveness, defined by an increase of cardiac output > 15% after fluid expansion (ΔCO-FE > 15%, gold-standard test)

SECONDARY OUTCOMES:
Diagnostic accuracy of the SAV mean and the ΔPeak for the diagnosis of fluid responsiveness | after abdominal compression, 30 minutes to 4 hours after baseline
  Diagnostic accuracy of the SAV mean and the ΔPeak for the diagnosis of fluid responsiveness, defined by an increase of cardiac output > 15% after fluid expansion (ΔCO-FE > 15%, gold-standard test) in preterm infants.
  Comparison of the diagnostic accuracy of these tests.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie CRAMAREGEAS, Principal Investigator — Bordeaux hospital University
Locations (1):
- Bordeaux Hospital University, Bordeaux, France